CLINICAL TRIAL: NCT06664047
Title: Radiological and Clinical Outcomes of Over-the-Top ACL Reconstruction vs. Anteromedial ACL Reconstruction With Additional Lateral Extraarticular Tenodesis: A Prospectively Randomized Controlled Trial
Brief Title: Over-the-Top vs. Anteromedial ACLR With Lateral Extraarticular Tenodesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Enejd Veizi, MD, Assistant Professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TADEB-1-24-645
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Tear
Keywords: Anterior cruciate ligament rupture; Over-the-top reconstruction; Lateral extra-articular tenodesis
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Prospectively Randomized Controlled Trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OTT ACLR (Active Comparator): Patients in this group will undergo a reconstruction with the OTT technique which includes an intra-articular component and an extra-articular one, functioning as a LET.
  Interventions: Procedure: OTT ACLR
- ACLR LET (Active Comparator): Patients in this group will undergo a reconstruction with the conventional ACL technique accompanied by a routine LET, obtained from the iliotibial band.
  Interventions: Procedure: ACLR LET

INTERVENTIONS:
Procedure: OTT ACLR — Patients in this group will undergo a reconstruction with the OTT technique which includes an intra-articular component and an extra-articular one, functioning as a LET.
  Arms: OTT ACLR
Procedure: ACLR LET — Patients in this group will undergo a reconstruction with the conventional ACL technique accompanied by a routine LET, obtained from the iliotibial band.
  Arms: ACLR LET

SUMMARY:
This study aims to compare the over-the-top (OTT) anterior cruciate ligament (ACL) reconstruction (ACL-R) technique with the anteromedial ACL-R + lateral extraarticular tenodesis (LET). It aims to provide valuable insights into two different surgical approaches aimed at enhancing knee stability. The over-the-top ACL-R technique, which involves routing the graft over the posterior aspect of the lateral femoral condyle, is known for its simplicity and ability to preserve the anatomical footprint of the ACL. Although a non-anatomical reconstruction, the OTT technique has shown comparable clinical results and good return to sports (RTS) ratios when compared to the conventional ACLR alone. It is also favored in revision surgeries or when there is difficulty accessing the femoral tunnel through conventional approaches. However, concerns regarding its ability to fully restore rotational stability persist, especially in high-demand athletes.

In contrast, the anteromedial portal technique for ACL-R, combined with LET, has gained popularity due to its effectiveness in controlling both anterior tibial translation and rotational instability. LET augments the intra-articular reconstruction by providing additional restraint against pivot shifts, which can be critical in patients with high-risk profiles for re-injury, such as those participating in pivoting sports. Comparing these two approaches in terms of clinical outcomes, graft integrity, rotational control, and return-to-sport rates with a prospectively randomized controlled trial will help clarify their roles in contemporary ACL surgery and could guide surgeons in choosing the most appropriate method based on patient-specific factors.

DETAILED DESCRIPTION:
Anterior cruciate ligament reconstruction (ACLR) is one of the most commonly performed procedures in orthopedic sports medicine, aimed at restoring knee stability, facilitating return to activities, and preventing secondary injuries to the cartilage and menisci. Improved understanding of knee joint anatomy and biomechanics has led to advancements in surgical techniques, and modern 'anatomic' techniques have shown favorable outcomes in most patients. However, despite technical advancements, ACL reconstruction techniques still fail to fully restore normal knee biomechanics, particularly with regard to tibial rotation, leaving some patients with residual instability. Additionally, the rate of return to high-level sports has been reported as low as 63% at two years.

Residual anterolateral subluxation, as measured by the pivot shift test, is a clinical indicator of internal rotation laxity and is associated with poor outcomes and low patient satisfaction. Such altered kinematics may contribute further to the development of osteoarthritis (OA). The inability of traditional ACLR to reliably restore normal tibial rotational kinematics could be one reason for this outcome.

Lateral extra-articular tenodesis (LET) is performed alongside ACLR to control anterolateral rotational instability in knees with ACL deficiency. Recent studies have shown that this procedure reduces the risk of ACL graft re-rupture, better restores knee joint kinematics, and improves return-to-sport rates. ACLR and LET procedures are now routinely performed in many centers.

The over-the-top (OTT) ACL reconstruction technique involves passing the graft over the superomedial edge of the lateral femoral condyle and securing it to the lateral femoral cortex. The proposed advantages of this technique include its safety, ease of use, reproducibility, low cost, and compatibility with all graft types and fixation methods. Additionally, the OTT technique can be used to reinforce ACL remnants, thus minimizing technical challenges encountered during anatomic reconstruction procedures. These challenges include difficulty visualizing the femoral placement, mismatches between tibial and femoral tunnels, reliance on clock-face systems for femoral tunnel positioning, and instrument impingement during excessive knee flexion.

Currently, there is limited literature comparing the outcomes of OTT and anatomic ACLR techniques, and no studies compare the OTT and ACLR + LET procedures.

The aim of this study is to compare the clinical and radiological outcomes, as well as return-to-sport rates, between patients undergoing the Over-the-Top ACL Reconstruction technique and those undergoing the Anteromedial ACL Reconstruction technique with Lateral Extra-Articular Tenodesis.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an isolated anterior cruciate ligament (ACL) tear (isolated ligament injury).
* Age between 18 and 50 years.
* No previous history of surgery on the same knee.
* MRI and CT scans performed at the end of the first postoperative year.

Exclusion Criteria:

* Presence of additional ligamentous injury (e.g., posterior cruciate ligament or collateral ligament) along with the ACL tear.
* Incomplete clinical scores.
* History of previous surgery on the same knee.
* Presence or history of infection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Re-rupture | Postoperative 1.st year
  Re-rupture prevalence detected on MRI (yes/no)
Tibial tunnel widening | Postoperative 1.st year
  Tibial tunnel diameter measured at the widest point on axial CT scans (number, mm)
Tegner Activity Scale | Postoperative 1.st year
  minimum value:0, maximum value 10, higher values mean better outcome
Knee Score ve Knee Injury & Osteoarthritis Outcome (KOOS) | Postoperative 1.st year
  minimum value:0, maximum value 100, higher values mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Enejd Veizi, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lucidi GA, Roberti di Sarsina T, Zaffagnini S. Editorial Commentary: The Number One Cause of Anterior Cruciate Ligament Reconstruction Graft Failure Is a Misplaced Femoral Tunnel: Over-the-Top Technique Plus Lateral Extra-Articular Tenodesis Is Recommended. Arthroscopy. 2024 Feb;40(2):435-437. doi: 10.1016/j.arthro.2023.07.021. PMID 38296446
- [Background] Zaffagnini S, Lucidi GA, Macchiarola L, Agostinone P, Neri MP, Marcacci M, Grassi A. The 25-year experience of over-the-top ACL reconstruction plus extra-articular lateral tenodesis with hamstring tendon grafts: the story so far. J Exp Orthop. 2023 Apr 1;10(1):36. doi: 10.1186/s40634-023-00599-8. PMID 37005946
- [Background] Kamei G, Nakamae A, Nakata K, Nekomoto A, Tsuji S, Hashiguchi N, Ishikawa M, Adachi N. Comparison of clinical outcomes between anterior cruciate ligament reconstruction with over-the-top route procedure and anatomic single-bundle reconstruction in pediatric patients. J Pediatr Orthop B. 2023 Mar 1;32(2):178-184. doi: 10.1097/BPB.0000000000001008. Epub 2023 Dec 15. PMID 36700965
- [Background] Bonanzinga T, Grassi A, Altomare D, Lucidi GA, Macchiarola L, Zaffagnini S, Marcacci M. High return to sport rate and few re-ruptures at long term in professional footballers after anterior cruciate ligament reconstruction with hamstrings. Knee Surg Sports Traumatol Arthrosc. 2022 Nov;30(11):3681-3688. doi: 10.1007/s00167-022-06944-1. Epub 2022 Apr 22. PMID 35451640